CLINICAL TRIAL: NCT01274221
Title: A Phase 3b, Randomized, Double-blind, Multicenter, Placebo Controlled, Dose Optimization, Crossover, Analog Classroom, Safety and Efficacy Study of SPD489 in Adolescent Subjects Aged 13-17 Years With Attention-Deficit/Hyperactivity Disorder (ADHD))
Brief Title: Safety and Efficacy of SPD489 in Adolescent Subjects Aged 13-17 Years With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Cancellation was not safety related but a shift in study priorities for Shire.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-321
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- SPD489 (Active Comparator)
  Interventions: Drug: SPD489

INTERVENTIONS:
Drug: SPD489 — 1 capsule per day throughout the open-label treatment phase and for one week of the double-blind crossover phase
  Other Names: Vyvanse, Lisdexamfetamine dimesylate, LDX
  Arms: SPD489
Other: Placebo — 1 capsule per day for one week of the double-blind crossover phase
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of SPD489 compared to placebo in adolescent subjects (13-17 years of age inclusive) with ADHD in the analog classroom setting based on the Permanent Product Measure of Performance (PERMP) total score assessed across 2, 4, 9, 13, 14, and 15 hours post-dose on the last day of each double-blind crossover period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or female, 13-17 years of age inclusive, at the time of consent.
2. The parent/LAR must be available at approximately 7:00 AM (±2 hours) to dispense the dose of investigational product for the study duration.
3. Subject, who is a female, must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test and a negative urine pregnancy test and agree to comply with any applicable contraceptive requirements of the protocol.
4. Subject meets the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation.
5. Subject has an Attention Deficit/Hyperactivity Disorder Rating Scale-Fourth Edition (ADHD-RS-IV) total score ≥28.
6. Subject is functioning at an age-appropriate level intellectually.
7. Subject is able to swallow a capsule.

Exclusion Criteria:

1. Subject has a current, controlled (with medications prohibited in this study) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any significant comorbid Axis II disorder or significant Axis I disorder (such as post traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, depressive or anxiety disorder) or other symptomatic manifestations that, in the opinion of the examining clinician, will contraindicate treatment with SPD489 or confound efficacy or safety assessments.
2. Subject has a documented history of aggressive behavior serious enough to preclude participation in regular classroom activities, as determined by the Investigator. Oppositional defiant disorder is not exclusionary.
3. Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently, demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator
4. Subject is underweight.
5. Subject is significantly overweight.
6. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject.
7. Subject has a history of seizures (other than infantile febrile seizures), a chronic or current tic disorder, a current diagnosis, and/or a known family history of Tourette's Disorder. Subject has a history of tics that are judged by the Investigator to be exclusionary.
8. Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place him/her at increased vulnerability to the sympathomimetic effects of a stimulant drug.
9. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
10. Subject has any clinically significant electrocardiogram (ECG) or clinically significant laboratory abnormality.
11. Subject has current abnormal thyroid function. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
12. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
13. Subject has failed to respond to 1 or more adequate courses (dose and duration) of amphetamine therapy.
14. Subject has a history of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria.
15. Subject has a positive urine drug result (with the exception of subject's current stimulant therapy, if any).
16. Subject has taken another investigational product or has taken part in a clinical study within 30 days prior to the Screening visit.
17. Subject has previously been screened for this study or has participated in any other SPD489/NRP104 clinical studies.
18. Subject has glaucoma.
19. Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
20. Subject is female and is pregnant or lactating.
21. Subject is well controlled on his/her current ADHD medication with acceptable tolerability.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-03-06 (Estimated); Primary Completion 2011-05-04 (Estimated); Study Completion 2011-05-04 (Estimated)

PRIMARY OUTCOMES:
Permanent Product Measure of Performance (PERMP) Total Score | 7 Days

SECONDARY OUTCOMES:
Attention Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Total Score | 7 Days
Conners' Parent Rating Scale - Revised (CPRS-R) Total Score | 7 Days
Clinical Global Impressions - Global Improvement (CGI-I) Rating Scale Score | 7 Days
Vital Signs (includes oral or tympanic temperature, sitting blood pressure, pulse and respiratory rate) and Body Height and Weight | Baseline, Weeks 7, 14, 21, 28, 35 and 42
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Weeks 7, 14, 21, 28, 35 and 42

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- United States (6):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Ltd., Houston, Texas
  - John M. Turnbow, MD, PA, Lubbock, Texas